CLINICAL TRIAL: NCT02772159
Title: A Single-Dose, Fixed-Sequence, Two-Period Study to Evaluate the Absorption, Distribution, Metabolism, Excretion of TD-4208 Following an IV Infusion and an Oral Dose of [14C]-Labeled TD-4208 in Healthy Male Subjects
Brief Title: TD-4208 Absorption, Distribution, Metabolism and Excretion (ADME) Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0130
Record Dates: First submitted 2015-06-10; First posted 2016-05-13 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; ADME; Healthy Normal Males; Phase 1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Population (Experimental): One dose each of treatments A: [14C] TD-4208 20 μg IV administered in a fasted state over 30 minutes. B: [14C] TD-4208 200 μg oral solution administered in a fasted state.
  Interventions: Drug: TD-4208

INTERVENTIONS:
Drug: TD-4208 — One dose each of treatments A: [14C] TD-4208 20 μg IV administered in a fasted state over 30 minutes. B: [14C] TD-4208 200 μg oral solution administered in a fasted state.
  Other Names: revefenacin

SUMMARY:
The purpose of this study is to evaluate the absorption, distribution, metabolism and excretion of an investigational medication used to treat chronic obstructive pulmonary disease (COPD). The study drug will be tested in 6 healthy normal males. Dosing will include a single dose of study drug administered via an IV Infusion and an Oral Dose. There will be a 28 day washout period between each of the 2 dosing routes.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, two-period study in up to 12 healthy male subjects. The present study is designed to fully characterize the rates and routes of elimination of TD 4208 using radiolabeled drug administered via the oral and IV route. This study will provide information regarding the metabolic fate of TD 4208, the need for evaluation of potential drug-drug interactions, the need for studies in special populations and the absolute oral bioavailability of TD-4208. The results from this study will allow a comprehensive comparison between animal and human routes of elimination and metabolic profiles of TD 4208.

This study will be conducted in a small number of healthy male subjects (up to n=12) to minimize the number of individuals exposed to radioactivity. Each subject will receive the following treatments: Treatment A (Period 1): 20 μg IV infusion of [14C] TD-4208 administered in a fasted state over 30 minutes. Treatment B (Period 2): 200 μg oral solution of [14C] TD-4208 administered in a fasted state. Blood, urine, feces, and vomitus (if applicable) will be collected until the subject is released during Periods 1 and 2. In Periods 1 and 2, subjects may remain in the clinical research unit for a maximum of 15 days. Between the dosing in periods 1 and 2, there will be washout intervals of at least 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a body mass index 19 to 32 kg/m2, inclusive, and weigh at least 55 kg.
2. Subject has normal blood pressure (BP) and heart rate (HR), measured after resting seated or supine for approximately 5 minutes. Normal BP is defined as 90 to 140 mm Hg systolic and 50 to 90 mm Hg diastolic. Normal HR is defined as 40 to 99 beats per minute.
3. Subject is negative for hepatitis B, hepatitis C, and HIV antibodies.
4. Subject has no clinically relevant abnormalities as determined by the investigator in the results of Screening or Day -1 laboratory evaluations.

Exclusion Criteria:

1. Subject has any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas]).
2. Subject has participated in another clinical trial of an investigational drug (or medical device) within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to Screening, or are currently participating in another trial of an investigational drug (or medical device).
3. Subject has a known hypersensitivity towards medications similar to TD-4208 or excipients contained in TD-4208.
4. Subject has previously participated in a trial for TD-4208.
5. Subject regularly works with ionizing radiation or radioactive material.
6. Subject has been exposed to ionizing radiations, within 1 year prior to the start of the study, as external irradiation (radiological examination including CT scan excluding dental radiography) or internal radiation (diagnostic nuclear medicine procedure) or have participated in a radiolabeled study in the last 12 months.
7. Subject has had exposure to external and/or internal radiotherapy with open (i.e., nuclear medicine) and sealed sources (i.e., brachytherapy) within the last 12 months.
8. Subject, who, for any reason, is deemed by the investigator to be inappropriate for this study or have any condition which would confound or interfere with the evaluation of the safety, tolerability, PK of the investigational drug or prevent compliance with the study protocol.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
[14C] total radioactivity in urine and reported as the recovery in urine as a percentage of the administered dose | up to 336 hours
[14C] total radioactivity in feces and reported as the recovery in feces as a percentage of the administered dose | up to 336 hours

SECONDARY OUTCOMES:
Whole blood concentrations of total radioactivity | up to 336 hours
Plasma concentrations of total radioactivity | up to 336 hours
Plasma concentrations of TD-4208 | up to 336 hours
Plasma concentrations of THRX-195518 | up to 336 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma, US, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No